CLINICAL TRIAL: NCT01863784
Title: An Open-Label Study to Evaluate the Pharmacokinetics of Multiple Oral Doses of 30 mg JNJ-38518168 in Subjects With Mild and Moderate Hepatic Impairment Compared With Subjects With Normal Hepatic Function
Brief Title: A Study to Evaluate the Pharmacokinetics of JNJ-38518168 in Patients With Mild and Moderate Hepatic Impairment Compared With Patients With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101336; 38518168ARA1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Mild and moderate hepatic impairment; Normal hepatic function; Pharmacokinetics; JNJ-38518168
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-38518168 (Experimental)
  Interventions: Drug: JNJ-38518168

INTERVENTIONS:
Drug: JNJ-38518168 — All participants will receive JNJ-38518168 30 mg tablet once daily from Day 1 to Day 14.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (what the body does to the study medication) of JNJ-38518168 at approximately steady-state (stable medication levels) after administration of multiple oral 30 mg doses of JNJ-38518168 to participants with mild or moderate hepatic (liver) impairment (abnormal function) compared with participants with normal hepatic function.

DETAILED DESCRIPTION:
This is an open-label (both [participants and investigator] know what treatment participants will receive) and multicenter study. The study consists of 3 phases: a screening phase (approximately 3 weeks), a treatment phase (from day -2 [2 days before the administration of study medication] to Day 18), and an end-of-study phase (7 to 10 days after the last dose of study medication). Approximately 24 participants (participants with mild hepatic impairment, moderate hepatic impairment, and normal liver function) will receive JNJ-38518168 for 14 days. Hepatic impairment will be evaluated according to Child-Pugh score. It consists of 5 clinical measures (amount of ascites [an abnormal accumulation of fluid in the abdomen], total bilirubin [mg/dL], albumin [g/dL], international normalized ratio, and degree of encephalopathy [abnormal functioning of the brain]). Each is scored from 0 (less severity) to 3 (highest severity). Total Child-Pugh score is the sum of all subscores and is graded as: mild (5-6 points), moderate (7-9 points), and severe (10-15 points). Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, vital signs, body weight, physical examination, and 12-lead electrocardiogram which will be monitored at various timepoints throughout the study. The total duration of study participation for each participant is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have normal liver function for the normal hepatic function group
* Have mild or moderate liver diseases as defined by the Child-Pugh Classification and be clinically stable overall for the mild or moderate liver disease groups
* Doses of drugs used to treat other illnesses or conditions related to liver disease must be stable for at least 4 weeks before the first dose of study medication with the exception of thyroid replacement hormone, in which case the dose must be stable for 3 months before the first dose of study medication. Doses of these drugs must also be stable during the course of the study
* If an illness with a fever occurs within one week of the start of dosing, dosing must be postponed until the body temperature is normal for at least 72 hours
* Participants must agree to use one of the contraception methods defined in the protocol

Exclusion criteria:

* Hepatic insufficiency secondary to autoimmune hepatitis or obstructive liver disease
* Allergy to heparin or history of heparin-induced thrombocytopenia
* All participants must have a negative human immunodeficiency virus test. Participants with normal liver function must test negative for hepatitis B and hepatitis C
* Severe ascites (an abnormal accumulation of fluid in the abdomen) or severe pleural effusion (fluid around the lungs)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of JNJ-38518168 at approximately steady-state after multiple doses | Day 14 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, and 96 hours])
Area under the plasma concentration-time curve of JNJ-38518168 at approximately steady-state after multiple doses | Day 14 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, and 96 hours])
Time to reach the maximum observed plasma of JNJ-38518168 at approximately steady-state after multiple doses | Day 14 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, and 96 hours])
Apparent clearance of JNJ-38518168 at approximately steady-state after multiple doses | Day 14 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, and 96 hours])

SECONDARY OUTCOMES:
Maximum observed plasma concentration of JNJ-38518168 after single dose | Day 1 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours])
Area under the plasma concentration-time curve of JNJ-38518168 after single dose | Day 1 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours])
Time to reach the maximum observed plasma of JNJ-38518168 after single dose | Day 1 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours])
Urine concentration-time data of JNJ-38518168 after single dose | Day 1 (predose, postdose [1, 2, 3, 4, 5, 6, 7, 8, 12, and 24 hours])
Plasma protein binding of JNJ-38518168 | Day 1 (postdose [4 hours]) and Day 14 (predose, postdose [4 hours])
Number of participants with adverse events | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Orlando, Florida
  - Knoxville, Tennessee
  - San Antonio, Texas